CLINICAL TRIAL: NCT02221401
Title: Bioequivalence of a 2.5 mg Linagliptin / 1000 mg Metformin Fixed-dose Combination Tablet Compared With Single Linagliptin 2.5 mg and Metformin 1000 mg Tablets Administered Together in Healthy Male and Female Volunteers (an Open-label, Randomised, Single Dose, Two-way Crossover, Phase I Trial)
Brief Title: Bioequivalence of a Linagliptin / Metformin Fixed-dose Combination (FDC) Tablet Compared With Single Linagliptin and Metformin Tablets Administered Together in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.1
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Metformin

ARMS (2):
- Treatment A (FDC) (Experimental)
  Interventions: Drug: Linagliptin/Metformin FDC
- Treatment B (single agents) (Active Comparator)
  Interventions: Drug: Linagliptin; Drug: Metformin

INTERVENTIONS:
Drug: Linagliptin/Metformin FDC
  Arms: Treatment A (FDC)
Drug: Linagliptin
  Arms: Treatment B (single agents)
Drug: Metformin
  Arms: Treatment B (single agents)

SUMMARY:
Study to demonstrate bioequivalence of a 2.5 mg linagliptin/1000 mg metformin fixed-dose combination (FDC) tablet compared with single tablets of linagliptin 2.5 mg and metformin 1000 mg administered together.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women according to the following criteria: based upon a complete medical history, including physical examination, vital signs (Blood pressure (BP), Pulse Rate (PR)), 12-lead ECG, clinical laboratory tests
2. Age 18 to 55 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Surgery of the gastrointestinal tract (except appendectomy)
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
6. History of relevant orthostatic hypotension, fainting spells or blackouts
7. Chronic or relevant acute infections
8. History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
9. Intake of drugs within 1 month or less than 10 half-lives of the respective drug prior to first study drug administration
10. Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
11. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes daily)
12. Alcohol abuse (average consumption of more than 20 g/day in women and 30 g/day in men)
13. Drug abuse
14. Blood donation (more than 100 mL within 4 weeks before Day 1 of Visit 2)
15. Any laboratory value outside the reference range of clinical relevance
16. Inability to comply with dietary regimen of trial site

    For female subjects of childbearing potential only:
17. Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 2 months after study completion
18. No adequate contraception during the study and until 1 month after study completion, e.g. not any of the following: implants, injectables, combined hormonal contraceptives, hormonal intrauterine device, sexual abstinence for at least 1 month prior to first study drug administration, vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilization (including hysterectomy). Women who did not have a vasectomised partner, were not sexually abstinent or surgically sterile were asked to use an additional barrier method (e.g. condom).
19. Lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
AUC0-72 (area under the concentration-time curve of linagliptin in plasma over the time interval from 0 to 72 h) | up to 72 hours
Cmax (maximum measured concentration of the analyte in plasma) | up to 72 hours
AUC0-∞ (area under the concentration-time curve of metformin in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of linagliptin in plasma over the time interval from 0 extrapolated to infinity) | up to 72 hours
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 72 hours
%AUCtz-∞ (percentage of AUCtz-∞ obtained by extrapolation) | up to 72 hours
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval t1 to t2) | up to 72 hours
tmax (time from dosing until maximum concentration of the analyte in plasma) | up to 72 hours
λz (terminal elimination rate constant in plasma) | up to 72 hours
t1/2 (terminal half-life of the analyte in plasma) | up to 72 hours
MRTpo (mean residence time of the analyte in the body after peroral administration) | up to 72 hours
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 72 hours
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 72 hours
Number of subjects with clinically significant findings in vital signs | up to 7 days after last drug administration
  blood pressure, pulse rate
Number of subjects with clinically significant findings in 12-lead electrocardiogram (ECG) | up to 7 days after last drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 7 days after last drug administration
Number of subjects with adverse events | up to 7 days after last drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 7 days after last drug administration